CLINICAL TRIAL: NCT06826807
Title: Hepatic Elastography-Enhanced Lifestyle Modification in Patients With Metabolic Dysfunction-Associated Steatotic Liver Disease: A Randomized Controlled Trial
Brief Title: Hepatic Elastography-Enhanced Lifestyle Modification in MASLD
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Phunchai Charatcharoenwitthaya, Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SI 009/2025
Record Dates: First submitted 2025-01-28; First posted 2025-02-14 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Transient Elastography; MASLD; BMI; Metabolic Syndrome; NAFLD; Insulin Resistance; Cardiovascular Diseases
Keywords: Lifestyle modification; MASLD; transient elastography
MeSH Terms: conditions — Metabolic Syndrome; Non-alcoholic Fatty Liver Disease; Insulin Resistance; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: The intervention group will undergo regular hepatic elastography monitoring to assess liver fat composition and receive feedback to encourage dietary modifications and increased physical activity. The control group will receive standard care without elastography monitoring.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Active Comparator: Regular hepatic elastography monitoring to encourage dietary modifi (Experimental): • MASLD patient will undergo regular hepatic elastography monitoring to assess liver fat composition and receive feedback to encourage dietary modifications and increased physical activity.
  Interventions: Other: Regular monitoring with transient elastography
- No Intervention: Placebo comparator: standard care (counselling for dietary modifications and increa (No Intervention): The control group will receive standard care (counselling for dietary modifications and increased physical activity) without elastography monitoring.

INTERVENTIONS:
Other: Regular monitoring with transient elastography — MASLD patients were received their liver fat and fibrosis status regularly using transient elastography
  Arms: Experimental: Active Comparator: Regular hepatic elastography monitoring to encourage dietary modifi

SUMMARY:
The 2022 National Health Survey in Thailand revealed a substantial rise in obesity and metabolic dysfunction-associated steatotic liver disease (MASLD). The prevalence of MASLD was 19.7%, with higher rates observed in individuals with metabolic syndrome and diabetes. Effective management of MASLD primarily involves lifestyle modifications, including dietary adjustments and increased physical activity. Evidence suggests that patients unaware of their liver fibrosis status are less likely to adhere to these interventions. This study aims to evaluate the impact of hepatic elastography monitoring on lifestyle modification adherence and health outcomes in patients with MASLD over 48 weeks.

DETAILED DESCRIPTION:
The 2022 health survey of Thai adults (aged ≥18 years) reported an obesity prevalence of 44.9% (40.3% in males, 49.2% in females), a significant increase over past decades. Obesity is a major contributing factor to the rising incidence of MASLD, previously termed nonalcoholic fatty liver disease (NAFLD). MASLD is defined as fatty liver disease occurring in individuals consuming less than 140 grams of alcohol per week for females or less than 210 grams per week for males, alongside clinical features of metabolic dysfunction.

Among 18,588 surveyed individuals, the prevalence of MASLD was 19.7% (20.9% in males, 18.6% in females), with notably higher rates of 43.5% in those with abdominal obesity and 35.6% in individuals with diabetes. Significant associations were observed between MASLD and factors such as age, sex, physical activity, smoking, and metabolic abnormalities, including overweight, abdominal obesity, elevated triglycerides, diabetes, hypertension, and low HDL cholesterol levels.

MASLD is closely linked to insulin resistance, a critical risk factor for cardiovascular disease. Current guidelines emphasize weight loss through dietary control and exercise to reduce hepatic fat accumulation, inflammation, and fibrosis, while improving metabolic parameters such as blood glucose, lipid profiles, and insulin sensitivity. Behavioral and environmental factors, including high-calorie diets and sedentary lifestyles, contribute to the pathogenesis of MASLD by promoting insulin resistance and hepatic fat accumulation, leading to oxidative stress, inflammation, and fibrosis, thereby increasing the risks of cirrhosis and hepatocellular carcinoma.

A recent study highlighted that 59.2% of MASLD patients were unaware of their liver fat and fibrosis status. Lack of awareness was associated with poor adherence to lifestyle modifications, particularly in obese individuals (BMI > 30 kg/m²). This randomized controlled trial investigates the effect of hepatic elastography monitoring on lifestyle changes, hepatic steatosis, metabolic parameters, and anthropometry, compared to standard care over a 48-week period.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be diagnosed with MASLD according to the diagnostic criteria outlined in the multi-society Delphi consensus statement on new fatty liver disease nomenclature 2023, with evidence of hepatic steatosis and alcohol consumption of less than 140 grams per week for females or less than 210 grams per week for males, along with at least one clinical characteristic of metabolic syndrome.
2. Participants must be at least 18 years old and less than 80 years old at the time of enrollment.

Exclusion Criteria:

1. Individuals diagnosed with other chronic liver diseases, including hepatitis B or C, autoimmune hepatitis, Wilson's disease, liver cancer, hemochromatosis, or liver cirrhosis.
2. Individuals diagnosed with conditions that may influence MASLD, such as HIV, chronic inflammatory diseases, or connective tissue disorders.
3. Individuals taking medications known to promote fatty liver disease, such as amiodarone, steroids, methotrexate, hormonal medications, or immunosuppressants.
4. Individuals who have previously taken medications known to impact fatty liver disease, including vitamin E, pioglitazone, GLP-1 receptor agonists, or SGLT2 inhibitors.
5. Participants intending to join weight loss programs or undergo bariatric surgery for obesity treatment.
6. Individuals with severe chronic diseases presenting symptoms during physical activity, such as coronary artery disease, chronic obstructive pulmonary disease, or severe osteoarthritis, which may exacerbate their condition.
7. Patients with contraindications to undergoing MRI examinations, such as claustrophobia or incompatible body implants or materials.
8. Women who are pregnant.
9. Individuals who do not provide formal consent to participate in the research project.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in non-invasive marker magnetic resonance imaging-estimated proton density fat fraction (MRI-PDFF) (%) | 48 weeks
  Hepatic fat content assessed by MRI-PDFF (%)

SECONDARY OUTCOMES:
Change from baseline in non-invasive liver fibrosis marker | 48 weeks
  Liver fibrosis assessed by magnetic resonance elastography (kPa)
Change from baseline in markers of liver injury | 48 weeks
  Alanine aminotransferase (ALT) (U/L), aspartate aminotransferase (AST) (U/L), and gamma glutamyl transferase (GGT) (U/L).
Change from baseline in markers of glycemic control | 48 weeks
  Fasting blood glucose (mg/dL)
Change from baseline in Hemoglobin A1C (%) | 48 weeks
  Hemoglobin A1C (%)
Change from baseline in lipoproteins | 48 weeks
  To compare changes in total cholesterol, triglyceride, HDL-cholesterol, and LDL-Total cholesterol (mg/dL), Triglycerides (TG) (mg/dL), high density lipoprotein cholesterol (HDL-C) (mg/dL), Non-HDL-C (mg/dL), and low-density lipoprotein cholesterol (LDL-C) (mg/dL)
Change from baseline in body fat composition assessed by Bioelectrical Impedance Analysis | 48 weeks
  Body fat percentage assessed by Bioelectrical Impedance Analysis
Change from baseline in muscle mass assessed by Bioelectrical Impedance Analysis | 48 weeks
  Muscle mass in kilograms assessed by Bioelectrical Impedance Analysis
Change from baseline in visceral fat assessed by Bioelectrical Impedance Analysis | 48 weeks
  Visceral fat rate assessed by Bioelectrical Impedance Analysis
Change from baseline in wieght in kilograms assessed by Bioelectrical Impedance Analysis | 48 weeks
  Body wieght in kilograms assessed by Bioelectrical Impedance Analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkoknoi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sheka AC, Adeyi O, Thompson J, Hameed B, Crawford PA, Ikramuddin S. Nonalcoholic Steatohepatitis: A Review. JAMA. 2020 Mar 24;323(12):1175-1183. doi: 10.1001/jama.2020.2298. PMID 32207804
- [Background] Koolhaas CM, van Rooij FJ, Cepeda M, Tiemeier H, Franco OH, Schoufour JD. Physical activity derived from questionnaires and wrist-worn accelerometers: comparability and the role of demographic, lifestyle, and health factors among a population-based sample of older adults. Clin Epidemiol. 2017 Dec 18;10:1-16. doi: 10.2147/CLEP.S147613. eCollection 2018. PMID 29296097
- [Background] Joo JH, Kim HJ, Park EC, Jang SI. Association between sitting time and non-alcoholic fatty live disease in South Korean population: a cross-sectional study. Lipids Health Dis. 2020 Sep 23;19(1):212. doi: 10.1186/s12944-020-01385-6. PMID 32967678
- [Background] Mansour-Ghanaei R, Mansour-Ghanaei F, Naghipour M, Joukar F. The Lifestyle Characteristics in Non-Alcoholic Fatty Liver Disease in the PERSIAN Guilan Cohort Study. Open Access Maced J Med Sci. 2019 Sep 14;7(19):3313-3318. doi: 10.3889/oamjms.2019.647. eCollection 2019 Oct 15. PMID 31949537
- [Background] Rinella ME, Neuschwander-Tetri BA, Siddiqui MS, Abdelmalek MF, Caldwell S, Barb D, Kleiner DE, Loomba R. AASLD Practice Guidance on the clinical assessment and management of nonalcoholic fatty liver disease. Hepatology. 2023 May 1;77(5):1797-1835. doi: 10.1097/HEP.0000000000000323. Epub 2023 Mar 17. No abstract available. PMID 36727674
- [Background] Akuta N, Kawamura Y, Arase Y, Suzuki F, Sezaki H, Hosaka T, Kobayashi M, Kobayashi M, Saitoh S, Suzuki Y, Ikeda K, Kumada H. Relationships between Genetic Variations of PNPLA3, TM6SF2 and Histological Features of Nonalcoholic Fatty Liver Disease in Japan. Gut Liver. 2016 May 23;10(3):437-45. doi: 10.5009/gnl15163. PMID 26610348
- [Background] Carrieri P, Mourad A, Marcellin F, Trylesinski A, Calleja JL, Protopopescu C, Lazarus JV. Knowledge of liver fibrosis stage among adults with NAFLD/NASH improves adherence to lifestyle changes. Liver Int. 2022 May;42(5):984-994. doi: 10.1111/liv.15209. Epub 2022 Mar 7. PMID 35220673
- [Background] Rinella ME, Lazarus JV, Ratziu V, Francque SM, Sanyal AJ, Kanwal F, Romero D, Abdelmalek MF, Anstee QM, Arab JP, Arrese M, Bataller R, Beuers U, Boursier J, Bugianesi E, Byrne CD, Castro Narro GE, Chowdhury A, Cortez-Pinto H, Cryer DR, Cusi K, El-Kassas M, Klein S, Eskridge W, Fan J, Gawrieh S, Guy CD, Harrison SA, Kim SU, Koot BG, Korenjak M, Kowdley KV, Lacaille F, Loomba R, Mitchell-Thain R, Morgan TR, Powell EE, Roden M, Romero-Gomez M, Silva M, Singh SP, Sookoian SC, Spearman CW, Tiniakos D, Valenti L, Vos MB, Wong VW, Xanthakos S, Yilmaz Y, Younossi Z, Hobbs A, Villota-Rivas M, Newsome PN; NAFLD Nomenclature consensus group. A multisociety Delphi consensus statement on new fatty liver disease nomenclature. Hepatology. 2023 Dec 1;78(6):1966-1986. doi: 10.1097/HEP.0000000000000520. Epub 2023 Jun 24. PMID 37363821
- [Background] Schneider CV, Zandvakili I, Thaiss CA, Schneider KM. Physical activity is associated with reduced risk of liver disease in the prospective UK Biobank cohort. JHEP Rep. 2021 Mar 2;3(3):100263. doi: 10.1016/j.jhepr.2021.100263. eCollection 2021 Jun. PMID 33898961
- [Background] Stens NA, Bakker EA, Manas A, Buffart LM, Ortega FB, Lee DC, Thompson PD, Thijssen DHJ, Eijsvogels TMH. Relationship of Daily Step Counts to All-Cause Mortality and Cardiovascular Events. J Am Coll Cardiol. 2023 Oct 10;82(15):1483-1494. doi: 10.1016/j.jacc.2023.07.029. Epub 2023 Sep 6. PMID 37676198
- [Background] Boeckmans J, Gatzios A, Schattenberg JM, Koek GH, Rodrigues RM, Vanhaecke T. PNPLA3 I148M and response to treatment for hepatic steatosis: A systematic review. Liver Int. 2023 May;43(5):975-988. doi: 10.1111/liv.15533. Epub 2023 Feb 16. PMID 36719059
- [Background] Trepo E, Romeo S, Zucman-Rossi J, Nahon P. PNPLA3 gene in liver diseases. J Hepatol. 2016 Aug;65(2):399-412. doi: 10.1016/j.jhep.2016.03.011. Epub 2016 Mar 30. PMID 27038645
- [Background] Romeo S, Kozlitina J, Xing C, Pertsemlidis A, Cox D, Pennacchio LA, Boerwinkle E, Cohen JC, Hobbs HH. Genetic variation in PNPLA3 confers susceptibility to nonalcoholic fatty liver disease. Nat Genet. 2008 Dec;40(12):1461-5. doi: 10.1038/ng.257. Epub 2008 Sep 25. PMID 18820647
- [Background] Anstee QM, Day CP. The Genetics of Nonalcoholic Fatty Liver Disease: Spotlight on PNPLA3 and TM6SF2. Semin Liver Dis. 2015 Aug;35(3):270-90. doi: 10.1055/s-0035-1562947. Epub 2015 Sep 17. PMID 26378644
- [Background] Maximos M, Bril F, Portillo Sanchez P, Lomonaco R, Orsak B, Biernacki D, Suman A, Weber M, Cusi K. The role of liver fat and insulin resistance as determinants of plasma aminotransferase elevation in nonalcoholic fatty liver disease. Hepatology. 2015 Jan;61(1):153-60. doi: 10.1002/hep.27395. Epub 2014 Nov 25. PMID 25145475
- [Background] European Association For The Study Of The Liver. Corrigendum to 'EASL recommendations on treatment of hepatitis C: Final update of the series' [J Hepatol 73 (2020) 1170-1218]. J Hepatol. 2023 Feb;78(2):452. doi: 10.1016/j.jhep.2022.10.006. Epub 2022 Dec 1. No abstract available. PMID 36464532
- [Background] Zelber-Sagi S, Nitzan-Kaluski D, Goldsmith R, Webb M, Zvibel I, Goldiner I, Blendis L, Halpern Z, Oren R. Role of leisure-time physical activity in nonalcoholic fatty liver disease: a population-based study. Hepatology. 2008 Dec;48(6):1791-8. doi: 10.1002/hep.22525. PMID 18972405
- [Background] St George A, Bauman A, Johnston A, Farrell G, Chey T, George J. Independent effects of physical activity in patients with nonalcoholic fatty liver disease. Hepatology. 2009 Jul;50(1):68-76. doi: 10.1002/hep.22940. PMID 19444870
- [Background] Gerber L, Otgonsuren M, Mishra A, Escheik C, Birerdinc A, Stepanova M, Younossi ZM. Non-alcoholic fatty liver disease (NAFLD) is associated with low level of physical activity: a population-based study. Aliment Pharmacol Ther. 2012 Oct;36(8):772-81. doi: 10.1111/apt.12038. Epub 2012 Sep 8. PMID 22958053
- [Background] Hallsworth K, Thoma C, Moore S, Ploetz T, Anstee QM, Taylor R, Day CP, Trenell MI. Non-alcoholic fatty liver disease is associated with higher levels of objectively measured sedentary behaviour and lower levels of physical activity than matched healthy controls. Frontline Gastroenterol. 2015 Jan;6(1):44-51. doi: 10.1136/flgastro-2014-100432. Epub 2014 Jun 30. PMID 25580206
- [Background] Koutoukidis DA, Koshiaris C, Henry JA, Noreik M, Morris E, Manoharan I, Tudor K, Bodenham E, Dunnigan A, Jebb SA, Aveyard P. The effect of the magnitude of weight loss on non-alcoholic fatty liver disease: A systematic review and meta-analysis. Metabolism. 2021 Feb;115:154455. doi: 10.1016/j.metabol.2020.154455. Epub 2020 Nov 29. PMID 33259835
- [Background] Romero-Gomez M, Zelber-Sagi S, Trenell M. Treatment of NAFLD with diet, physical activity and exercise. J Hepatol. 2017 Oct;67(4):829-846. doi: 10.1016/j.jhep.2017.05.016. Epub 2017 May 23. PMID 28545937
- [Background] Shen J, Wong GL, Chan HL, Chan RS, Chan HY, Chu WC, Cheung BH, Yeung DK, Li LS, Sea MM, Woo J, Wong VW. PNPLA3 gene polymorphism and response to lifestyle modification in patients with nonalcoholic fatty liver disease. J Gastroenterol Hepatol. 2015 Jan;30(1):139-46. doi: 10.1111/jgh.12656. PMID 25040896
- [Background] Hernaez R, Lazo M, Bonekamp S, Kamel I, Brancati FL, Guallar E, Clark JM. Diagnostic accuracy and reliability of ultrasonography for the detection of fatty liver: a meta-analysis. Hepatology. 2011 Sep 2;54(3):1082-1090. doi: 10.1002/hep.24452. PMID 21618575
- [Background] Stine JG, Munaganuru N, Barnard A, Wang JL, Kaulback K, Argo CK, Singh S, Fowler KJ, Sirlin CB, Loomba R. Change in MRI-PDFF and Histologic Response in Patients With Nonalcoholic Steatohepatitis: A Systematic Review and Meta-Analysis. Clin Gastroenterol Hepatol. 2021 Nov;19(11):2274-2283.e5. doi: 10.1016/j.cgh.2020.08.061. Epub 2020 Aug 31. PMID 32882428
- [Background] Karlas T, Petroff D, Sasso M, Fan JG, Mi YQ, de Ledinghen V, Kumar M, Lupsor-Platon M, Han KH, Cardoso AC, Ferraioli G, Chan WK, Wong VW, Myers RP, Chayama K, Friedrich-Rust M, Beaugrand M, Shen F, Hiriart JB, Sarin SK, Badea R, Jung KS, Marcellin P, Filice C, Mahadeva S, Wong GL, Crotty P, Masaki K, Bojunga J, Bedossa P, Keim V, Wiegand J. Individual patient data meta-analysis of controlled attenuation parameter (CAP) technology for assessing steatosis. J Hepatol. 2017 May;66(5):1022-1030. doi: 10.1016/j.jhep.2016.12.022. Epub 2016 Dec 28. PMID 28039099
- [Background] Saint-Maurice PF, Troiano RP, Berrigan D, Kraus WE, Matthews CE. Volume of Light Versus Moderate-to-Vigorous Physical Activity: Similar Benefits for All-Cause Mortality? J Am Heart Assoc. 2018 Apr 2;7(7):e008815. doi: 10.1161/JAHA.118.008815. PMID 29610219
- [Background] Kwak MS, Kim D, Chung GE, Kim W, Kim JS. The preventive effect of sustained physical activity on incident nonalcoholic fatty liver disease. Liver Int. 2017 Jun;37(6):919-926. doi: 10.1111/liv.13332. Epub 2016 Dec 24. PMID 27917585
- [Background] Asada F, Nomura T, Hosui A, Kubota M. Influence of increased physical activity without body weight loss on hepatic inflammation in patients with nonalcoholic fatty liver disease. Environ Health Prev Med. 2020 Jun 10;25(1):18. doi: 10.1186/s12199-020-00857-6. PMID 32522147
- [Background] Kistler KD, Brunt EM, Clark JM, Diehl AM, Sallis JF, Schwimmer JB; NASH CRN Research Group. Physical activity recommendations, exercise intensity, and histological severity of nonalcoholic fatty liver disease. Am J Gastroenterol. 2011 Mar;106(3):460-8; quiz 469. doi: 10.1038/ajg.2010.488. Epub 2011 Jan 4. PMID 21206486
- [Background] Bird SR, Hawley JA. Update on the effects of physical activity on insulin sensitivity in humans. BMJ Open Sport Exerc Med. 2017 Mar 1;2(1):e000143. doi: 10.1136/bmjsem-2016-000143. eCollection 2016. PMID 28879026
- [Background] Kim D, Murag S, Cholankeril G, Cheung A, Harrison SA, Younossi ZM, Ahmed A. Physical Activity, Measured Objectively, Is Associated With Lower Mortality in Patients With Nonalcoholic Fatty Liver Disease. Clin Gastroenterol Hepatol. 2021 Jun;19(6):1240-1247.e5. doi: 10.1016/j.cgh.2020.07.023. Epub 2020 Jul 16. PMID 32683103
- [Background] LaMonte MJ, Lewis CE, Buchner DM, Evenson KR, Rillamas-Sun E, Di C, Lee IM, Bellettiere J, Stefanick ML, Eaton CB, Howard BV, Bird C, LaCroix AZ. Both Light Intensity and Moderate-to-Vigorous Physical Activity Measured by Accelerometry Are Favorably Associated With Cardiometabolic Risk Factors in Older Women: The Objective Physical Activity and Cardiovascular Health (OPACH) Study. J Am Heart Assoc. 2017 Oct 17;6(10):e007064. doi: 10.1161/JAHA.117.007064. PMID 29042429
- [Background] White T, Westgate K, Wareham NJ, Brage S. Estimation of Physical Activity Energy Expenditure during Free-Living from Wrist Accelerometry in UK Adults. PLoS One. 2016 Dec 9;11(12):e0167472. doi: 10.1371/journal.pone.0167472. eCollection 2016. PMID 27936024
- [Background] Jeon CY, Lokken RP, Hu FB, van Dam RM. Physical activity of moderate intensity and risk of type 2 diabetes: a systematic review. Diabetes Care. 2007 Mar;30(3):744-52. doi: 10.2337/dc06-1842. PMID 17327354
- [Background] Goodpaster BH, Katsiaras A, Kelley DE. Enhanced fat oxidation through physical activity is associated with improvements in insulin sensitivity in obesity. Diabetes. 2003 Sep;52(9):2191-7. doi: 10.2337/diabetes.52.9.2191. PMID 12941756
- [Background] Engin A. The Definition and Prevalence of Obesity and Metabolic Syndrome. Adv Exp Med Biol. 2017;960:1-17. doi: 10.1007/978-3-319-48382-5_1. PMID 28585193
- [Background] Ekstedt M, Nasr P, Kechagias S. Natural History of NAFLD/NASH. Curr Hepatol Rep. 2017;16(4):391-397. doi: 10.1007/s11901-017-0378-2. Epub 2017 Nov 13. PMID 29984130
- [Background] Younossi ZM, Koenig AB, Abdelatif D, Fazel Y, Henry L, Wymer M. Global epidemiology of nonalcoholic fatty liver disease-Meta-analytic assessment of prevalence, incidence, and outcomes. Hepatology. 2016 Jul;64(1):73-84. doi: 10.1002/hep.28431. Epub 2016 Feb 22. PMID 26707365